CLINICAL TRIAL: NCT04733274
Title: Patient and Healthcare Professional Views on Genetic/Genomic Information and Testing
Status: Active, not recruiting | Type: Observational
Sponsor: Boston College (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Andrew Dwyer, Associate Professor, Boston College
Other Study IDs: 18.081.01
Record Dates: First submitted 2021-01-25; First posted 2021-02-02 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Hypogonadism, Hypogonadotropic; Kallmann Syndrome
MeSH Terms: conditions — Hypogonadism; Kallmann Syndrome

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Technologic advances (i.e. next generation sequencing technologies and novel bioinformatics approaches) have been drivers of scientific discovery and have deepened our understanding of the genetics and genomics of health and disease. In parallel, the falling cost of sequencing has led to screening moving from specialty clinics into the primary care setting. However, our ability to help patients and families understand these technologies and related genetic health literacy issues lag behind. These factors pose a number of questions and challenges for clinicians including: how can we best present complex genetic/genomic information to patients to ensure that patients understand the information and can make informed decisions? What are the specific information and support needs of patients and families to be able to make decisions that are in line with their values? In collaboration with investigators from the Harvard Reproductive Endocrine Sciences Center at the Massachusetts General Hospital, this project broadly aims to examine patient understanding and factors affecting decisions surrounding genetic testing. Using the paradigm of a rare genetic disorder (isolated gonadotropin releasing hormone [GnRH] deficiency - hypogonadotropic hypogonadism/Kallmann syndrome [HH/KS]) we will examine the views and perspectives of patients and healthcare professionals alike regarding genetic/genomic information and testing with the intention of identifying patient-centered responses to these unmet needs and challenges.

DETAILED DESCRIPTION:
The focus of this study is to better understand perspectives on genetic testing. The study will collect and analyze both quantitative and qualitative data form healthcare professionals as well as patients. Findings will be used to inform more person-centered approaches to genetic testing that will support high-quality decisions that are informed and aligned with patient values and preferences. To achieve this, the study has three specific aims.

Aim 1. Evaluate the understandability and acceptability of education materials (including information on genetic testing) co-created with patients.

Patient education materials will be created drawing on healthcare professionals expertise (i.e. content experts) and patients (i.e. lived experience). Quality of materials will be quantitatively measured using the gold standard Patient Education Materials Assessment Tool (PEMAT).

Aim 2. Identify the central elements for a patient decision aid using expert clinician opinion.

Healthcare professionals who are content experts in the field will be surveyed to determine key information for a proposed genetic testing decision aid. Quantitative findings will guide the content of a patient decision aid for genetic testing.

Aim 3. Explore patient needs for information and support related to genetic testing.

Qualitative focus groups with patients will be conducted and analyzed using thematic analysis. Findings will inform the development of a patient decision aid for genetic testing that is responsive to the aspects which matter most to patients.

ELIGIBILITY:
Inclusion Criteria:

1. self-identified as having been diagnosed with either normosmic hypogonadotropic hypogonadism (HH) or Kallmann syndrome (KS)
2. between the ages of 18-70 years
3. primary language is English/capable of responding to a written questionnaire in English
4. has lived in the United states for 5 years or longer
5. checking the opt-in electronic consent

Exclusion Criteria:

1. other diagnosis of hypogonadism i.e. Klinefelter syndrome, or adult-onset hypogonadotropic hypogonadism
2. outside the stated age range

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with either normosmic hypogonadotropic hypogonadism (HH) or Kallmann syndrome (KS)
Sampling Method: Non-Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the understandability and acceptability of education materials (including information on genetic testing) cocreated with patients | 1-hour post-test
  Patient Education Materials Assessment Tool (PEMAT): higher scores indicate materials that are more readily understood and actionable by patients
Identify the central elements for a patient decision aid using expert clinician opinion | baseline
  survey with Likert-type scale questions: higher scores indicate a perceived higher priority for respective items/topic matter
Explore patient needs for information and support related to genetic testing | baseline
  Qualitative focus group findings (thematic analysis) - open ended questions will probe the nature of experiences with genetic testing as well as perceived promoters and barriers to testing and sharing results with potentially at-risk blood relatives

SECONDARY OUTCOMES:
Compare face-to-face and virtual focus group formats | baseline
  similarities/differences in face-to-face vs. virtual focus groups - emergent themes form face-to-face and virtual focus groups will be compared to identify similarities/differences in the type and quantity of elicited codes

CONTACTS AND LOCATIONS:
Overall Officials: Andrew A Dwyer, PhD, Principal Investigator — Boston College
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston College, Chestnut Hill, Massachusetts

REFERENCES:
- [Background] Dwyer AA, Uveges M, Dockray S, Smith N. Advancing qualitative rare disease research methodology: a comparison of virtual and in-person focus group formats. Orphanet J Rare Dis. 2022 Sep 11;17(1):354. doi: 10.1186/s13023-022-02522-3. PMID 36089593
- [Result] Dwyer AA, Zeng Z, Lee CS. Validating online approaches for rare disease research using latent class mixture modeling. Orphanet J Rare Dis. 2021 May 10;16(1):209. doi: 10.1186/s13023-021-01827-z. PMID 33971926
- [Result] Dwyer AA, Uveges MK, Dockray S, Smith N. Exploring Rare Disease Patient Attitudes and Beliefs regarding Genetic Testing: Implications for Person-Centered Care. J Pers Med. 2022 Mar 16;12(3):477. doi: 10.3390/jpm12030477. PMID 35330476